CLINICAL TRIAL: NCT06373783
Title: Ultrasonographic Evaluation of the Efficacy of Subepithelial Connective Tissue Grafts Versus De-epithelized Gingival Graft in Root Coverage With Coronally Advanced Flap Technique
Brief Title: Ultrasonographic Evaluation of the Connective Tissue Grafts Obtained With Two Different Methods in Root Coverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Gizem Torumtay Cin, asistant prof., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/05
Record Dates: First submitted 2024-04-04; First posted 2024-04-18 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Gingival Recession, Localized
Keywords: Connective tissue graft; gingival recession; ultrasonography; de-epithelized gingival graft; tissue thickness; blood-flow velocity
MeSH Terms: conditions — Gingival Recession | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- de-epithelise (Active Comparator): In combination with Zuchelli's coronally positioned flap technique, gingival recession in the upper jaw premolar region was treated using a de-epithelialized gingival graft. The gingival graft was taken in a rectangular shape from the area located on the palatal side of the maxillary canine and the first molar tooth, and then it was de-epithelised with the help of a scalpel.
  Interventions: Procedure: de- epithelize gingival graft; Diagnostic Test: ultrasonography
- subepithelial (Active Comparator): In combination with Zuchelli's coronally positioned flap technique, gingival recession in the upper jaw premolar region was treated using a subepithelial gingival graft. Connective tissue taken from the upper jaw-palate region with a single incision technique was used.
  Interventions: Procedure: subepithelial connective tissue graft; Diagnostic Test: ultrasonography

INTERVENTIONS:
Procedure: subepithelial connective tissue graft — The area where the gingival recession occurred was prepared with the modified coronally positioned flap technique developed by Zuchelli. The subepithelial connective tissue graft was obtained in each patient using the single incision technique from the region between the mesial of the canine and the mesial of the first molar in the palate. Connective tissue dimensions were approximately 10x5x2 mm. The graft thickness was measured with an endodontic spreader from 3 points (mesial, buccal, and distal) and an electronic caliper during surgery.
  Arms: subepithelial
Procedure: de- epithelize gingival graft — The area where the gingival recession occurred was prepared with the modified coronally positioned flap technique developed by Zuchelli. A shallow horizontal incision was made at ≈3 mm apical from the gingival margin of the maxillary molar teeth using a number 15 scalpel blade. Subsequently, a parallel horizontal incision, at ≈ 4 mm apical from the first horizontal incision, was traced in conjunction with two vertical releasing incisions to delineate a rectangular area. Then, the uppermost epithelial layer was scraped off using a size 11 scalpel tip. The connective tissue graft to be taken from the palate area was 10x5x2 mm in size, and the graft thickness was measured with an endodontic spreader from 3 points (mesial, buccal, and distal) and electronic caliper during surgery.
  Arms: de-epithelise
Diagnostic Test: ultrasonography — Clinical parameter measurements (probing depth (PD), clinical attachment level (CAL), gingival recession depth and width, keratinized tissue width and height) were taken on the day of surgery, the 3rd days, the 14th days, the 1st month, the 3rd months and the 6th months.
  Ultrasonography measurements A 6-18 MHz intraoral probe was used in intraoral USG examinations. Sterile gel was applied to the intraoral probe and covered with a stretch film. Then, it was placed directly on the mucosal surface of the receiver site in the buccal area. Mucosal thickness was evaluated using the B-mode of the device, and vascularization was evaluated using the color doppler and pulsed wave doppler modes of the device. The following equation is used and calculated by US unit pulsatility index (PI) = (Vmax-Vmin) (Vmean) (Vmax is peak systolic flow velocity. Vmin is diastolic flow velocity and Vmean is mean flow velocity.) The mean PI values of each patient were measured.

SUMMARY:
Gingival recession is a clinical problem that increases with age and affects patient comfort. It is defined as the displacement of the gingival margin to a more apical position of the cementum-enamel border of the tooth.

Coronally advanced flap (CAF) or tunnel technique (TUN) with subepithelial connective tissue procedures have been reported to be the most predictable methods of single gingival recession treatments. The ultimate goal of these plastic periodontal surgical procedures is to close the exposed root surface and achieve optimum aesthetic results. The main indications for root coverage (RC) procedures are aesthetic concern, root hypersensitivity, prevention of cervical abrasion and root caries, improvement of restorative results, and facilitation of plaque control. The use of a subepithelial connective tissue graft (SCGT) combined with a coronally positioned flap is considered the gold standard by many authors for single gingival recession treatments.

De-epithelialization of free gingival grafts (DGG) has been proposed, especially when palatal tissue thickness is insufficient (≤2.5 mm) and larger graft size in the apico-coronal or mesio-distal directions is required. In this technique, the graft of the required width and length is separated from the lateral side of the palate, and then the 0.3-0.5 mm thick epithelial layer of the resulting graft is cut from the connective tissue layer.

Ultrasonography (USG) is based on the principle of recording data obtained as a result of ultrasound waves sent with the help of a probe hitting and reflecting on substances of different densities. This technique is widely used in medical practice. In dentistry, the USG method is used to measure the alveolar bone level and the dimensions of the periodontium to evaluate the gingival thickness. It also has functions to evaluate color power and color speed, as well as blood flow.

The study hypothesizes that combining SCGT and DGG with a coronally positioned flap could yield different clinical outcomes in patients with a single buccal gingival recession. This study aims to compare the clinical success of connective tissue grafts obtained by two different surgical methods in covering the root surface with ultrasonography (USG).

DETAILED DESCRIPTION:
The study was planned as a randomized controlled study. Patients with single Miller class 1 or 2 gingival recession who need root coverage surgery in the Department of Periodontology were included in the study. In combination with Zuchelli's coronally positioned flap technique, gingival recession in the upper jaw premolar region was treated using a de-epithelialized gingival graft or a subepithelial gingival graft. The subepithelial connective tissue graft was obtained in each patient using the single incision technique from the region between the mesial of the canine and the mesial of the first molar in the palate. Connective tissue dimensions were approximately 10 X 5 X 2 mm. Finally, the incision line was sutured with 5/0 synthetic, nonabsorbable, sterile monofilament suture. The de-epithelized gingival graft was taken in a rectangular shape from the area located on the palatal side of the maxillary canine and the first molar tooth, and then it was de-epithelized with the help of a scalpel. After the graft was stabilized to the recipient area with a 5-0 resorbable, sterile monofilament suture. The flap was repositioned and sutured with 5/0 synthetic, nonabsorbable, sterile monofilament suture.

Clinical measurements (probing depth (PD), clinical attachment level (CAL), gingival recession depth and width, keratinized tissue width and height) were taken on the day of surgery, the 3rd days, the 14th days, the 1st month, the 3rd months and the 6th months.

Patients were evaluated using an ultrasonography device ( MyLabtm Seven, Esaote, Genoa, Italy) at the Department of Oral and Maxillofacial Radiology.

USG measurements were performed on days 0, 3, 14, 30, 90, and 180 for buccal tissue thickness and tissue vascularization by an oral and maxillofacial radiologist with at least six years of experience. A 6-8 MHZ intraoral probe was used in intraoral USG examinations. Steril gel was applied to the intraoral probe and covered with stretch film. Then, it was placed directly on the buccal mucosal surface. Mucosal thickness was evaluated using the B-mode of the device, and vascularization was evaluated using the color Doppler and pulsed wave Doppler modes of the device. mean pulsatility index (PI) values of each patient were calculated and considered for statistical analysis.

The power analysis of the study was performed for sample size calculation. In the power analysis, when α = 0.05, β = 0.40, 1-β: 0.80, the number of regions to be included in the study was determined as 20 for each group. The sample size was calculated with a statistical program.

The data obtained from the study is the 22. version of SPSS. (SPSS Inc., Chicago, IL) descriptive analysis, means and standard deviations were calculated for all clinical effects, and USG measurements. Repeated measures analysis of variance was used for intragroup comparisons before and after treatment. The normality of data distributions of the groups was measured with the Kolmogorov-Smirnov test. In the comparison of groups, an independent groups t-test was used if the data distributions were normal, and Mann Whitney U test was used if the data distribution was not normal. The significance value was taken as p<00.5.m (G*Power; Universitat, Dusseldorf, Germany).

ELIGIBILITY:
Inclusion Criteria:

* Patients with single Miller class 1 or 2 gingival recession who have undergone root coverage surgery.
* 18 to 65 years old
* non-smoker and non-alcoholic.
* Patients who have good oral hygiene and whose inflammation can be controlled (FMPS <25%, FMBS <25%, probing depth ≤ 3mm, and bleeding on probing <10%)
* Those who have no previous history of periodontal surgery in the operation area

Exclusion Criteria:

* Active smokers
* pregnancy and lactation
* Continuation of gingival trauma due to false tooth brushing
* Presence of severe tooth malposition
* Those with systemic diseases that may affect wound healing after periodontal surgery
* Individuals who cannot maintain oral hygiene

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-03-16 (Actual)

PRIMARY OUTCOMES:
tissue thickness | at baseline before operation, on days 3,14, 30, 90,180
  tissue thickness was measured with B-Mod mod of ultrasonography device

SECONDARY OUTCOMES:
pulsatility index | at baseline before operation, on days 3,14,30,90,180
  pulsatility index was measured with Doppler-mode of ultrasonography device.

CONTACTS AND LOCATIONS:
Overall Officials: GİZEM TORUMTAY CİN, assist prof., Principal Investigator — PAMUKKALE UNIVERSITY FACULTY of DENTISTIRY
Locations (1):
- Pamukkale University of the Dentistry, Denizli, Turkey (Türkiye)